CLINICAL TRIAL: NCT01620840
Title: Lacosamid-i.v.-Register
Acronym: LCM
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Ulrich Stephani, Prof. Dr. med. Ulrich Stephani, University Hospital Schleswig-Holstein
Other Study IDs: UCB-LCM-2011
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Epilepsy With Partial Onset Seizures With or Without Secondary Generalization
Keywords: oral administration of Lacosamide is not possible or adequate
MeSH Terms: interventions — Lacosamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lacosamid-i.v. treatment
  Interventions: Drug: Lacosamide 10mg/ml

INTERVENTIONS:
Drug: Lacosamide 10mg/ml — intravenous administration up to 10 days
  Other Names: VimpatⓇ

SUMMARY:
Lacosamide is a new antiepileptic drug (AED) marketed as Vimpat with three different formulations, tablets, oral syrup and a solution for intravenous infusion. Lacosamide is approved as adjunctive therapy in epilepsy patients with partial onset seizures with or without secondary generalization. The i.v. solution is used in patients in which oral administration is not possible or adequate. Bioequivalence with oral tablets and safety could be demonstrated in healthy volunteers and in patients switched from tablets to Lacosamide i.v. solution. A recently published study demonstrates the feasibility of single loading doses up to 300 mg. The aim of this Lacosamide i.v. registry is to collect systematically data on the safety, tolerability and administration procedures when Lacosmide i.v. is used in routine daily clinical practice, mainly in hospitals. These data will help treating physicians to optimize the use of Lacosamide i.v. in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* before any data are collected for any patient in this registry an ehtical committee must be notified of the registry and written data consent must be properly executed and documented

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated with Lacosamide i.v.-solution in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2011-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Stephani, Prof.Dr.med., Principal Investigator — University hospital Schleswig-Holstein, Germany
Locations (1):
- Universitätsklinikum Schleswig-Holstein, Campus Kiel, Klinik für Neurologie, Kiel, Schleswig-Holstein, Germany